CLINICAL TRIAL: NCT02800720
Title: Meditation Awareness Training for the Treatment of Fibromyalgia Syndrome: A Randomised Controlled Trial
Brief Title: Meditation Awareness Training for the Treatment of Fibromyalgia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham Trent University (Other)
Responsible Party: Principal Investigator, William Van Gordon, Principal Investigator, Nottingham Trent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTU-MATFMS
Record Dates: First submitted 2016-06-06; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia Syndromey
MeSH Terms: conditions — Fibromyalgia | interventions — Cognitive Behavioral Therapy; Population Groups

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Meditation Awareness Training (Experimental): Target Intervention Arm:
  8-week meditation intervention
  Interventions: Behavioral: Meditation Awareness Training
- Cognitive Behavioural Therapy for Groups (Active Comparator): Active Comparator Arm:
  8-week CBT-based intervention
  Interventions: Behavioral: Cognitive Behavioral Therapy for Groups

INTERVENTIONS:
Behavioral: Meditation Awareness Training — 8 Week Meditation Intervention
  Arms: Meditation Awareness Training
Behavioral: Cognitive Behavioral Therapy for Groups — 8 week intervention based on Cognitive Behavioral Theory
  Arms: Cognitive Behavioural Therapy for Groups

SUMMARY:
A Randomised Controlled Trial to evaluate the effectiveness of a Second-Generation Mindfulness-Based Intervention known as Meditation Awareness Training (MAT) for treating fibromyalgia syndrome.

DETAILED DESCRIPTION:
Background: Fibromyalgia syndrome (FMS) is a chronic pain disorder that frequently leads to poor quality of life. The need for more effective FMS treatments has prompted empirical investigations into the applications of mindfulness for treating the condition. However, studies have predominantly focused on first-generation mindfulness-based interventions (FG-MBIs). To date, a randomised controlled trial (RCT) assessing the effectiveness of a second-generation mindfulness-based intervention (SG-MBI) for treating FMS has not been undertaken. SG-MBIs are distinct from FG-MBIs because they are overtly spiritual in nature and employ (i) a greater range of (normally secularised) meditative/spiritual techniques, (ii) ethics as a key component of the taught programme, and (iii) an instructor training programme that typically requires several years of supervised mindfulness practice.

Aims: To evaluate the effectiveness of Meditation Awareness Training (MAT) - an SG-MBI - for treating FMS.

Method: Adults with FMS will receive MAT or an active control intervention known as Cognitive-Behavioural Therapy for Groups. Assessments will be performed at pre-intervention, post-intervention, and follow-up phases.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of fibromyalgia syndrome
* Aged between 18 and 65 years
* Able to read and write using the English language
* Available to complete an eight-week intervention and six-month follow-up assessment

Exclusion Criteria:

* Currently undergoing formal psychotherapy
* Changes in psychopharmacology type or dosage one-month prior to intervention
* Currently practicing mindfulness or meditation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2012-11; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire | 8 weeks
  Scale Reference: Bennett, Friend, Jones, Ward, Han & Ross (2009)
Short Form McGill Pain Questionnaire | 8 weeks
  Scale Reference: Melzack (1987)
Pittsburgh Sleep Quality Index | 8 weeks
  Scale Reference: Buysse, Reynolds Monk, Berman, & Kupfer (1989)
Depression Anxiety and Stress Scale | 8 weeks
  Scale Reference: Lovibond & Lovibond (1995)

CONTACTS AND LOCATIONS:
Overall Officials: William Van Gordon, Principal Investigator — Nottingham Trent University

REFERENCES:
- Available data/document: Embedded Qualitative Study — http://link.springer.com/article/10.1007/s12671-015-0458-8